CLINICAL TRIAL: NCT01765582
Title: Steam (Sequencing Triplet With Avastin and Maintenance): FOLFOXIRI/Bevacizumab Regimens (Concurrent and Sequential) vs. FOLFOX/Bevacizumab in First-Line Metastatic Colorectal Cancer
Brief Title: Sequential and Concurrent FOLFOXIRI/Bevacizumab Regimens Versus FOLFOX/Bevacizumab in First-Line Metastatic Colorectal Cancer
Acronym: STEAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28442
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Capecitabine; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Concurrent FOLFOXIRI + Bevacizumab (Experimental): Participants will receive concurrent FOLFOXIRI along with 5 mg/kg of bevacizumab with treatment cycle of 2 weeks during first 4 month induction phase (plus optional 2 months of induction for participants who exhibit good response and tolerate the regimen) followed by administration of 5-FU with bevacizumab or capecitabine with bevacizumab as per investigator's discretion in maintenance phase. Following progression on first-line therapy (PD1), bevacizumab (dose equivalent, 2.5 mg/kg/week) will be administered as second-line therapy in combination with fluoropyrimidine based chemotherapy at the investigator's discretion.
  Interventions: Drug: 5-fluorouracil; Drug: bevacizumab; Drug: capecitabine; Drug: irinotecan; Drug: folinic acid; Drug: oxaliplatin
- Arm B: Sequential FOLFOXIRI + Bevacizumab (Experimental): Participants will receive alternating 4-week administrations of FOLFOX/bevacizumab and folinic acid (leucovorin), 5-FU, and irinotecan (FOLFIRI) /Bevacizumab with a treatment cycle of 2 weeks during first 4-month induction phase (plus optional 2 months of induction for participants who exhibit good response and tolerate the regimen) followed by administration of 5-FU with bevacizumab or capecitabine with bevacizumab as per investigator's discretion in maintenance phase. Following progression on first-line therapy (PD1), bevacizumab (dose equivalent, 2.5 mg/kg/week) will be administered as second-line therapy in combination with fluoropyrimidine based chemotherapy at the investigator's discretion.
  Interventions: Drug: 5-fluorouracil; Drug: bevacizumab; Drug: capecitabine; Drug: irinotecan; Drug: folinic acid; Drug: oxaliplatin
- Arm C: FOLFOX + Bevacizumab (Experimental): Participants will receive FOLFOX along with 5 mg/kg of bevacizumab with treatment cycle of 2 weeks during first 4-month induction phase (plus optional 2 months of induction for participants who exhibit good response and tolerate the regimen) followed by administration of 5-FU with bevacizumab or capecitabine with bevacizumab as per investigator's discretion in maintenance phase. Following progression on first-line therapy (PD1), bevacizumab (dose equivalent, 2.5 mg/kg/week) will be administered as second-line therapy in combination with fluoropyrimidine based chemotherapy at the investigator's discretion.
  Interventions: Drug: 5-fluorouracil; Drug: bevacizumab; Drug: capecitabine; Drug: folinic acid; Drug: oxaliplatin

INTERVENTIONS:
Drug: 5-fluorouracil — Participants in Arm A will receive 3200 milligrams per square meter (mg/m^2) by 48-hour continuous intravenous (IV) infusion every 2 weeks, during the 4-6 months' induction followed by maintenance therapy including bolus dose of 400 mg/m^2, followed by a 46-hour continuous infusion (2400 mg/m^2) every 2 weeks per investigator's discretion. Participants in Arm B and C will receive a bolus dose of 400 mg/m^2, followed by a 46-hour continuous infusion (2400 mg/m^2) every 2 weeks during the 4-6 months of induction and maintenance per investigator's discretion.
Drug: bevacizumab — Participants will receive 5 mg/kg IV every 2 weeks during the first 4-6 months induction phase, followed by 5 mg/kg IV every 2 weeks or 7.5 mg/kg IV every 3 weeks during maintenance therapy, and 2.5 mg/kg per week reinduction after disease progression.
  Other Names: Avastin
Drug: capecitabine — Participants will receive 1000 or 850 mg/kg orally twice daily as per investigator's discretion on Day 1 to 14, repeated every 3 weeks in maintenance phase.
  Other Names: Xeloda
Drug: irinotecan — Participants will receive IV infusion of 165 mg/m^2 over 1 hour every 2 weeks (Arm A) or IV infusion of 180 mg/m^2 over 1 hour in 2 x 2 weeks cycles alternating months (in Arm B), during 4-6 months induction phase.
  Arms: Arm A: Concurrent FOLFOXIRI + Bevacizumab; Arm B: Sequential FOLFOXIRI + Bevacizumab
Drug: folinic acid — Participants will receive IV infusion of 200 mg/m^² (Arm A) or 400 mg/m^2 (Arm B or C) over 2 hours every 2 weeks, during 4-6 months induction phase followed by IV infusion of 400 mg/m^2 in the maintenance therapy.
  Other Names: leucovorin
Drug: oxaliplatin — Participants will receive 85 mg/m^2 over 2 hours as IV infusion every 2 weeks (Arm A, C ) or 2 x 2 week cycles alternating months (Arm B), during 4-6 months induction phase .

SUMMARY:
This randomized, open-label, multicenter study will evaluate the efficacy and safety of folinic acid (leucovorin), 5-fluorouracil (5-FU), oxaliplatin, and irinotecan (FOLFOXIRI) / bevacizumab regimens (concurrent and sequential) versus folinic acid (leucovorin), 5-fluorouracil, and oxaliplatin (FOLFOX) / bevacizumab in first-line in participants with metastatic colorectal cancer. Participants will be randomized to receive bevacizumab 5 milligrams per kilogram (mg/kg) intravenously every 2 weeks with either concurrent or sequential FOLFOXIRI or with FOLFOX for 4 to 6 months of induction therapy, followed by maintenance therapy with bevacizumab plus either leucovorin/5-fluorouracil or capecitabine until disease progression occurs. After disease progression, participants will receive treatment with a fluoropyrimidine-based chemotherapy plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer with at least one measurable metastatic lesion by RECIST v 1.1, that is considered unresectable at baseline
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 if age less than (<) 71 years; ECOG status of 0 if age 71 to 75 years
* Adequate hematological, renal and liver function
* Participants with treated brain metastases are eligible for study participation; participants may not receive ongoing treatment with steroids at screening, anticonvulsants (at stable dose) are allowed
* Females of childbearing potential and males must agree to use effective contraception as defined by protocol during the treatment period and for at least 6 months after the last dose of study drug

Exclusion Criteria:

* Any prior treatment for metastatic colorectal cancer, except for use of palliative radiosensitizers
* Adjuvant chemotherapy for colorectal cancer completed < 12 months prior to study consent
* Sensory peripheral neuropathy greater than or equal to (>/=) Grade 2
* Evidence of Gilbert's Syndrome or homozygosity for the Uridine 5-diphospho-glucuronosyltransferase (UGT) 1A1*28 allele
* Positive for human immunodeficiency virus (HIV) infection
* Malignancies other than metastatic colorectal cancer within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent
* Radiotherapy to any site for any reason within 28 days prior to randomization, except for palliative radiotherapy to bone lesions within 14 days prior to randomization
* Clinically significant third-space fluid collections (e.g. ascites or pleural effusion) that cannot be controlled by drainage or other procedures prior to study entry
* Treatment with any other investigational agent, or participation in another investigational drug trial within 28 days prior to randomization
* Any disease or condition or laboratory finding giving reasonable suspicion of disease or condition that contraindicates the use of bevacizumab or puts the participant at high risk for treatment-related complications
* Inadequately controlled hypertension
* Clinically significant (that is [i.e.] active) cardiovascular disease (For example [e.g.] cerebrovascular accident or myocardial infarction within 6 months prior to randomization), unstable angina, congestive heart failure (New York Heart Association Class >/= II) or serious cardiac arrhythmia that is uncontrolled by medication or may interfere with the administration of the study treatment
* Known hypersensitivity to bevacizumab or any of its excipients or any other study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-01-23 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (45):
  - University of South Alabama; Mitchell Cancer Institute, Mobile, Alabama
  - Long Beach Memorial Medical Center; Oncology, Long Beach, California
  - LAC-USC Medical Center, Los Angeles, California
  - USC Norris Cancer Center, Los Angeles, California
  - Pacific Cancer Care - Monterey, Monterey, California
  - Sacramento Center for Hematolo, Sacramento, California
  - Pacific Cancer Care, Salinas, California
  - Kaiser Permanente - Franklin, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Fort Myers (Colonial Center Dr), Fort Myers, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Emory University Clinic, Atlanta, Georgia
  - Central Georgia Cancer Care PC, Macon, Georgia
  - Summit Cancer Care PC, Savannah, Georgia
  - Ingalls Memorial Hosp, Harvey, Illinois
  - Edward Cancer Center Naperville, Naperville, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Johns Hopkins Univ; Bunting Blaustein Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital; Cancer Care Center., Ann Arbor, Michigan
  - Karmanos Cancer Institute.., Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Southeast Nebraska Cancer Center;; Southeast Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Methodist Hospital; Cancer Center, Omaha, Nebraska
  - Dartmouth Hitchcock Med Center, Lebanon, New Hampshire
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - University of Oklahoma; Stephenson Oklahoma Canc Ctr, Oklahoma City, Oklahoma
  - Milton S. Hershey Medical Center; Penn State Cancer Inst., Hershey, Pennsylvania
  - Chattanooga Oncology and Hematology Associates, PC, Chattanooga, Tennessee
  - West Clinic, Germantown, Tennessee
  - Sarah Cannon Cancer Center and Research Institute, Nashville, Tennessee
  - UT Southwestern MC at Dallas, Dallas, Texas
  - Ctr for Cancer and Blood Disorders, Fort Worth, Texas
  - Scott and White Hospital; Cancer Center, Temple, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Seattle Cancer Care Alliance - Evergreen Health, Kirkland, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
  - Vince Lombardi Cancer Center, Green Bay, Wisconsin
  - Medical College of Wisconsin; Dept Froedtert Clin Can Ctr, Milwaukee, Wisconsin
  - Aurora Research Institute, Wauwatosa, Wisconsin
  - Cheyenne Oncology & Hematology Associates, Cheyenne, Wyoming

REFERENCES:
- [Derived] Cremolini C, Antoniotti C, Stein A, Bendell J, Gruenberger T, Rossini D, Masi G, Ongaro E, Hurwitz H, Falcone A, Schmoll HJ, Di Maio M. Individual Patient Data Meta-Analysis of FOLFOXIRI Plus Bevacizumab Versus Doublets Plus Bevacizumab as Initial Therapy of Unresectable Metastatic Colorectal Cancer. J Clin Oncol. 2020 Aug 20:JCO2001225. doi: 10.1200/JCO.20.01225. Online ahead of print. PMID 32816630
- [Derived] Hurwitz HI, Tan BR, Reeves JA, Xiong H, Somer B, Lenz HJ, Hochster HS, Scappaticci F, Palma JF, Price R, Lee JJ, Nicholas A, Sommer N, Bendell J. Phase II Randomized Trial of Sequential or Concurrent FOLFOXIRI-Bevacizumab Versus FOLFOX-Bevacizumab for Metastatic Colorectal Cancer (STEAM). Oncologist. 2019 Jul;24(7):921-932. doi: 10.1634/theoncologist.2018-0344. Epub 2018 Dec 14. PMID 30552157

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Concurrent FOLFOXIRI + Bevacizumab: Participants received concurrent FOLFOXIRI along with 5 mg/kg of bevacizumab with treatment cycle of 2 weeks during first 4 month induction phase (plus optional 2 months of induction for participants who exhibited good response and tolerated the regimen) followed by administration of 5-fluorouracil (5-FU) with bevacizumab or capecitabine with bevacizumab as per investigator's discretion in maintenance phase. Following progression on first-line therapy (PD1), bevacizumab (dose equivalent, 2.5 mg/kg/week) was administered as second-line therapy in combination with fluoropyrimidine based chemotherapy at the investigator's discretion.
- Arm B: Sequential FOLFOXIRI + Bevacizumab: Participants received alternating 4-week administrations of FOLFOX/bevacizumab and folinic acid (leucovorin), 5-FU, and irinotecan (FOLFIRI) /Bevacizumab with a treatment cycle of 2 weeks during first 4-month induction phase (plus optional 2 months of induction for participants who exhibited good response and tolerated the regimen) followed by administration of 5-FU with bevacizumab or capecitabine with bevacizumab as per investigator's discretion in maintenance phase. Following progression on first-line therapy (PD1), bevacizumab (dose equivalent, 2.5 mg/kg/week) was administered as second-line therapy in combination with fluoropyrimidine based chemotherapy at the investigator's discretion.
- Arm C: FOLFOX + Bevacizumab: Participants received FOLFOX along with 5 mg/kg of bevacizumab with treatment cycle of 2 weeks during first 4-month induction phase (plus optional 2 months of induction for participants who exhibited good response and tolerated the regimen) followed by administration of 5-FU with bevacizumab or capecitabine with bevacizumab as per investigator's discretion in maintenance phase. Following progression on first-line therapy (PD1), bevacizumab (dose equivalent, 2.5 mg/kg/week) was administered as second-line therapy in combination with fluoropyrimidine based chemotherapy at the investigator's discretion.
Period: Overall Study
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab
Started | 93 | 92 | 95
Completed | 0 | 0 | 0
Not Completed | 93 | 92 | 95
Not completed — Other | 3 | 6 | 9
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Death | 31 | 36 | 33
Not completed — Sponsor Decision | 46 | 42 | 42
Not completed — Withdrawal of Consent | 11 | 6 | 10

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population was defined as all randomized participants regardless of whether they received any dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Total
Number analyzed (Participants) | 93 | 92 | 95 | 280
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (11.53) | 56.0 (10.46) | 57.9 (9.86) | 56.7 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 36 | 118
  Male | 51 | 52 | 59 | 162

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response During First-Line Therapy (ORR1)
Description: ORR1 was the percentage of participants with complete response (CR) or partial response (PR) during first-line therapy as assessed by investigator according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v.1.1). CR was defined as disappearance of all extranodal target lesions and all pathological lymph nodes had to have decreased to <10 millimeter (mm) in short axis. PR was defined as at least a 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum diameters. ORR1 = CR + PR
Time Frame: Randomization up to disease progression during first-line therapy or death, whichever occurs first (up to approximately 3 years)
Population: ITT population was defined as all randomized participants regardless of whether they received any dose of study treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Arms A + B: Pooled FOLFOXIRI + Bevacizumab: This analysis set combines Arms A and B and represents participants who received either concurrent or sequential FOLFOXIRI with 5 mg/kg of bevacizumab during first 4-month induction phase (plus optional 2 months of induction for participants who exhibited good response and tolerated the regimen) followed by administration of 5-FU with bevacizumab or capecitabine with bevacizumab as per investigator's discretion in maintenance phase. Following progression on first-line therapy (PD1), bevacizumab (dose equivalent, 2.5 mg/kg/week) was administered as second-line therapy in combination with fluoropyrimidine based chemotherapy at the investigator's discretion.
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Arms A + B: Pooled FOLFOXIRI + Bevacizumab
Number analyzed (Participants) | 93 | 92 | 95 | 185
Percentage of participants | 72.0 | 72.8 | 62.1 | 72.4
Statistical Analysis 1: Comparison: Arm A: Concurrent FOLFOXIRI + Bevacizumab vs Arm C: FOLFOX + Bevacizumab; Stratified by extent of metastatic disease (liver-limited disease versus non liver-limited disease) and tumor location (right versus left) after correction post-randomization; Test type: Superiority or Other; p = 0.132, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.62, 90% CI 2-sided [0.96 to 2.71]

2. Primary Outcome: Progression-Free Survival During First-Line Therapy (PFS1)
Description: PFS1 was defined as time from randomization to the first occurrence of disease progression during first-line therapy, as assessed by the Investigator using RECIST v1.1, or death from any cause, whichever occurs first. Disease progression was defined as sum of longest diameters increased by at least 20% from the smallest value on study. The sum of longest diameters must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Arms A + B: Pooled FOLFOXIRI + Bevacizumab
Number analyzed (Participants) | 93 | 92 | 95 | 185
months | 11.86 [9.95 to 16.62] | 11.37 [9.20 to 13.34] | 9.46 [8.08 to 11.20] | 11.70 [10.35 to 13.34]
Statistical Analysis 1: Comparison: Arm C: FOLFOX + Bevacizumab vs Arms A + B: Pooled FOLFOXIRI + Bevacizumab; Stratified by extent of metastatic disease (liver-limited disease vs. non-liver-limited disease) and tumor location (right vs. left) after correction post-randomization; Test type: Superiority or Other; p = 0.005, Log Rank; Hazard Ratio (HR) = 0.68, 90% CI 2-sided [0.53 to 0.88]

3. Secondary Outcome: Time to PFS2
Description: Time to PFS2 was defined as time from randomization to the first occurrence of disease progression after reinduction of second-line therapy, as assessed by the Investigator using RECIST v1.1, or death from any cause, whichever occurs first. Disease progression was defined as sum of longest diameters increased by at least 20% from the smallest value on study. The sum of longest diameters must also demonstrate an absolute increase of at least 5mm.
Time Frame: Randomization up to disease progression during second-line therapy or death, whichever occurs first (up to approximately 3 years)
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Arms A + B: Pooled FOLFOXIRI + Bevacizumab
Number analyzed (Participants) | 24 | 30 | 29 | 54
months | 18.76 [13.63 to 24.31] | 13.17 [10.61 to 16.82] | 14.75 [11.01 to 16.13] | 15.08 [13.17 to 18.53]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Randomization until death due to any cause (up to approximately 3 years)
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Arms A + B: Pooled FOLFOXIRI + Bevacizumab
Number analyzed (Participants) | 93 | 92 | 95 | 185
months | 33.97 [23.69 to 33.97] | 28.32 [22.21 to NA] — N/A = NE = not evaluable: The value cannot be estimated because the curve representing the upper confidence limits for the survivor function lies above 0.5. | 30.65 [25.17 to 30.65] | 28.32 [23.75 to NA] — N/A = NE = not evaluable:The value cannot be estimated because the curve representing the upper confidence limits for the survivor function lies above 0.5.

5. Secondary Outcome: Proportion of Participants Who Underwent Liver Metastases Resections
Description: Reported here is the proportion of participants who underwent liver metastases resections calculated as follows: number of participants who underwent liver metastases resections divided by total number of participants in each arm.
Time Frame: Randomization up to approximately 3 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Arms A + B: Pooled FOLFOXIRI + Bevacizumab
Number analyzed (Participants) | 93 | 92 | 95 | 185
Proportion of participants | 0.17 [0.11 to 0.24] | 0.10 [0.05 to 0.15] | 0.08 [0.04 to 0.13] | 0.14 [0.09 to 0.18]

6. Secondary Outcome: Proportion of Participants Considered by the Investigator to be Unresectable on Study Enrollment Who Subsequently Underwent Attempted Curative Resections of Metastases
Description: The proportion of participants considered by the investigator to be unresectable at study enrollment who subsequently underwent attempted curative resections of metastases was calculated as follows: number of participants considered by the investigator to be unresectable at study enrollment who subsequently underwent attempted curative resections of metastases divided by total number of participants in each arm. This outcome represents a measure of the rate of conversion from unresectable to resectable disease.
Time Frame: Randomization up to approximately 3 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Arms A + B: Pooled FOLFOXIRI + Bevacizumab
Number analyzed (Participants) | 93 | 92 | 95 | 185
Proportion of participants | 0.24 [0.16 to 0.31] | 0.17 [0.11 to 0.24] | 0.14 [0.08 to 0.19] | 0.21 [0.16 to 0.25]

7. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Randomization up to approximately 3 years
Population: Safety population was defined as all randomized participants who received at least one partial or complete dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab | Arms A + B: Pooled FOLFOXIRI + Bevacizumab
Number analyzed (Participants) | 91 | 90 | 90 | 181
Percentage of participants | 100 | 98.9 | 100 | 99.4

ADVERSE EVENTS:
Time Frame: From baseline up to approximately 3 years.
Description: Safety population was defined as all randomized participants who received at least one partial or complete dose of study medication.
Arm/Group | Arm A: Concurrent FOLFOXIRI + Bevacizumab | Arm B: Sequential FOLFOXIRI + Bevacizumab | Arm C: FOLFOX + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 39/91 | 42/90 | 43/90
Other Adverse Events (participants affected / at risk) | 91/91 | 89/90 | 89/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Concurrent FOLFOXIRI + Bevacizumab (N=91) | Arm B: Sequential FOLFOXIRI + Bevacizumab (N=90) | Arm C: FOLFOX + Bevacizumab (N=90)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 5
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 3
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 3 | 5
Vomiting (Gastrointestinal disorders) | 3 | 0 | 4
Large intestine perforation (Gastrointestinal disorders) | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Medical device pain (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 5 | 1
Sepsis (Infections and infestations) | 1 | 2 | 4
Abdominal abscess (Infections and infestations) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Stoma site infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stoma obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 2
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder rupture (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 1
Air embolism (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Concurrent FOLFOXIRI + Bevacizumab (N=91) | Arm B: Sequential FOLFOXIRI + Bevacizumab (N=90) | Arm C: FOLFOX + Bevacizumab (N=90)
Neutropenia (Blood and lymphatic system disorders) | 42 | 43 | 29
Anaemia (Blood and lymphatic system disorders) | 16 | 17 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 12 | 9
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 5
Vision blurred (Eye disorders) | 17 | 9 | 7
Lacrimation increased (Eye disorders) | 4 | 8 | 7
Diarrhoea (Gastrointestinal disorders) | 73 | 65 | 49
Constipation (Gastrointestinal disorders) | 28 | 45 | 41
Abdominal pain (Gastrointestinal disorders) | 35 | 30 | 28
Dyspepsia (Gastrointestinal disorders) | 8 | 15 | 10
Abdominal pain upper (Gastrointestinal disorders) | 9 | 14 | 3
Flatulence (Gastrointestinal disorders) | 12 | 7 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 11 | 9
Abdominal distention (Gastrointestinal disorders) | 5 | 6 | 9
Haematochezia (Gastrointestinal disorders) | 8 | 3 | 5
Ascites (Gastrointestinal disorders) | 3 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 6 | 4 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 6 | 0
Nausea (Gastrointestinal disorders) | 59 | 64 | 53
Vomiting (Gastrointestinal disorders) | 33 | 36 | 24
Stomatitis (Gastrointestinal disorders) | 31 | 36 | 25
Haemorrhoids (Gastrointestinal disorders) | 7 | 11 | 12
Rectal haemorrhage (Gastrointestinal disorders) | 11 | 9 | 6
Oral pain (Gastrointestinal disorders) | 10 | 6 | 8
Proctalgia (Gastrointestinal disorders) | 8 | 4 | 5
Fatigue (General disorders) | 68 | 68 | 60
Temperature intolerance (General disorders) | 26 | 24 | 25
Mucosal inflammation (General disorders) | 16 | 16 | 14
Pyrexia (General disorders) | 16 | 10 | 15
Oedema peripheral (General disorders) | 10 | 11 | 6
Chills (General disorders) | 7 | 7 | 10
Pain (General disorders) | 4 | 11 | 9
Asthenia (General disorders) | 2 | 7 | 9
Chest pain (General disorders) | 6 | 4 | 1
Peripheral swelling (General disorders) | 6 | 3 | 2
Influenza like illness (General disorders) | 3 | 6 | 1
Oedema (General disorders) | 0 | 6 | 2
Hypersensitivity (Immune system disorders) | 2 | 2 | 6
Urinary tract infection (Infections and infestations) | 13 | 16 | 17
Upper respiratory tract infection (Infections and infestations) | 12 | 11 | 7
Sinusitis (Infections and infestations) | 6 | 11 | 2
Nasopharyngitis (Infections and infestations) | 4 | 3 | 6
Oral herpes (Infections and infestations) | 2 | 6 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 13 | 6 | 2
Fall (Injury, poisoning and procedural complications) | 5 | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 5 | 3 | 4
Weight decreased (Investigations) | 17 | 11 | 20
Neutrophil count decreased (Investigations) | 14 | 12 | 11
Aspartate aminotransferase increased (Investigations) | 6 | 7 | 4
White blood cell count decreased (Investigations) | 3 | 8 | 6
Blood alkaline phosphatase increased (Investigations) | 6 | 6 | 3
Blood bilirubin increased (Investigations) | 3 | 2 | 7
Platelet count decreased (Investigations) | 4 | 5 | 2
Deceased appetite (Metabolism and nutrition disorders) | 38 | 38 | 34
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 17 | 15
Dehydration (Metabolism and nutrition disorders) | 22 | 13 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 22 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 18 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 15 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 13 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1
Neuropathy peripheral (Nervous system disorders) | 33 | 32 | 32
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 30 | 36
Dysgeusia (Nervous system disorders) | 27 | 22 | 23
Headache (Nervous system disorders) | 26 | 29 | 17
Dizziness (Nervous system disorders) | 18 | 22 | 17
Paraesthesia (Nervous system disorders) | 9 | 12 | 14
Hypoaesthesia (Nervous system disorders) | 4 | 5 | 4
Insomnia (Psychiatric disorders) | 19 | 23 | 27
Anxiety (Psychiatric disorders) | 13 | 12 | 8
Depression (Psychiatric disorders) | 9 | 12 | 11
Proteinuria (Renal and urinary disorders) | 15 | 15 | 15
Dysuria (Renal and urinary disorders) | 3 | 4 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 | 30 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 30 | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 17 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 22 | 28 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 23 | 14
Rash (Skin and subcutaneous tissue disorders) | 9 | 17 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 11 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4 | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 4 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 | 6 | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 6 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Sinus operation (Surgical and medical procedures) | 2 | 5 | 1
Hypertension (Vascular disorders) | 35 | 36 | 24
Hot flush (Vascular disorders) | 10 | 6 | 3
Hypotension (Vascular disorders) | 7 | 2 | 10
Deep vein thrombosis (Vascular disorders) | 4 | 7 | 6
Embolism (Vascular disorders) | 1 | 5 | 0
Alanine aminotransferase increased (Investigations) | 6 | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 7

LIMITATIONS AND CAVEATS:
This trial was terminated on 12 November 2015, because the primary objective was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.